CLINICAL TRIAL: NCT04602923
Title: Comparison of Keratometric Change After Xen Gel Stent Implantation, Trabeculectomy, and Tube Shunts
Brief Title: Keratometric Change After XEN, Trabeculectomy and Tube Shunts
Acronym: Topo-XEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20.240
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Glaucoma Secondary; Glaucoma Eye
Keywords: Glaucoma drainage devices; Xen Gel Stent; Baerveldt glaucoma implant; Ahmed glaucoma implant; Trabeculectomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: 3 groups will be compared:
  * Group 1: 30 participants suffering from glaucoma who are candidates for XEN Gel Stent implantation
  * Group 2: 30 participants suffering from glaucoma who are candidates for trabeculectomy
  * Group 3: 30 participants suffering from glaucoma who are candidates for GDD implantation (BGI or AGV)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XEN Gel Stent implantation (Experimental): Participants suffering from glaucoma who are candidates for XEN Gel Stent implantation
  Interventions: Diagnostic Test: Corneal topography: OPD-Scan; Diagnostic Test: Corneal topography: Pentacam
- Trabeculectomy (Experimental): Participants suffering from glaucoma who are candidates for trabeculectomy
  Interventions: Diagnostic Test: Corneal topography: OPD-Scan; Diagnostic Test: Corneal topography: Pentacam
- GDD implantation (Experimental): Participants suffering from glaucoma who are candidates for GDD implantation (BGI or AGV)
  Interventions: Diagnostic Test: Corneal topography: OPD-Scan; Diagnostic Test: Corneal topography: Pentacam

INTERVENTIONS:
Diagnostic Test: Corneal topography: OPD-Scan — Corneal topography photography, taken by specular reflection (OPD-Scan) by measuring corneal curvature, thickness and topography.
Diagnostic Test: Corneal topography: Pentacam — Corneal topography photography, taken by Scheimpflug imaging (Pentacam) by measuring corneal curvature, thickness and topography.

SUMMARY:
The main goal of this study is to assess the severity of postoperative corneal astigmatism induced by implantation of the XEN Gel Stent compared to that induced by traditional filtering surgery (trabeculectomy and GDDs). Corneal astigmatism can be assessed using corneal topography, a non-invasive tool which provides an accurate estimate of corneal curvature in all meridians. To the best of our knowledge, no study has yet attempted to quantify the amount of astigmatism induced by the XEN Gel Stent.

DETAILED DESCRIPTION:
Following glaucoma surgery, patients often experience decreased visual acuity (VA) which can partly be explained by induced changes to the optical properties of the cornea. Corneal astigmatism can be assessed using corneal topography, a non-invasive tool which provides an accurate estimate of corneal curvature in all meridians. Obtained keratometric measures (termed K values) can allow clinicians to quantify the amount of astigmatism before and after surgical intervention.

Multiple studies have been previously published to evaluate induced postoperative astigmatism after trabeculectomy. However, only two studies have characterized the impact of GDDs on keratometric values. To the best of our knowledge, no study has yet attempted to quantify the amount of astigmatism induced by the XEN Gel Stent.

Assessing the impact of the XEN implant on corneal astigmatism is important to better characterize the expected course of postoperative visual rehabilitation, the impact of novel glaucoma devices on corneal properties and the predictability of refractive outcomes after XEN implantation. Compared to traditional filtering surgery, the XEN Gel Stent is inserted without opening the conjunctiva and is implanted further from the corneal limbus (5 mm). These factors may allow for a reduced amount of surgically induced corneal astigmatism.

We hypothesize that the XEN Gel Stent implantation induces less corneal astigmatism compared to traditional filtering surgery, such as the trabeculectomy and GDDs (BGI or AGV).

The main goal of this prospective interventional comparative study is to assess the severity of postoperative corneal astigmatism induced by implantation of the XEN Gel Stent compared to that induced by traditional filtering surgery (trabeculectomy and GDDs).

Secondary objectives are evaluation of visual acuity recovery as well as IOP reduction and other parameters between groups.

Glaucoma surgery (XEN Gel Stent, trabeculectomy or GDD implantation) will be performed by the ophthalmologists in charge of the study according to standard procedures. For each patient, the most appropriate type of glaucoma surgery will be recommended by the ophthalmologist regardless of patients' participation in the study, as dictated by the specific nature of their glaucoma and following current standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with an IOP above target and/or progressing on maximally tolerated medical therapy;
* Patients aged 18 years or older;
* Ability to provide informed consent;
* Ability to be followed for the entire duration of the study.

Exclusion Criteria:

* Patients less than 18 years old;
* Inability to provide informed consent;
* Inability to be followed for the entire duration of the study;
* Patients undergoing surgery combined with cataract extraction;
* Presence of severe dry eye disease;
* Presence of ocular comorbidities other than glaucoma, such as corneal or retinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Keratometric values (OPD-Scan) | Baseline, 2 months, 6 months, 12 months
  Change in simulated keratometric (K) values obtained by OPD-Scan between the indicated timepoints.
Keratometric values (Pentacam) | Baseline, 2 months, 6 months, 12 months
  Change in simulated keratometric (K) values obtained by Pentacam between the indicated timepoints.

SECONDARY OUTCOMES:
Best-corrected visual acuity change | Baseline, 2 months, 6 months, 12 months
  Evaluation of visual acuity change, measured using the Snellen chart.
Intraocular pressure change | Baseline, 2 months, 6 months, 12 months
  Evaluation of intraocular pressure control, measured using gold standard Goldmann applanation tonometry.
Visual field change change | Baseline, 6 months, 12 months
  Evaluation of visual field change. Visual field change will be calculated using the mean deviation (MD) values and pattern standard deviation (PSD) values measured using automated Humphrey 24-2 perimetry.
Retinal nerve fiber layer thickness change | Baseline, 6 months, 12 months
  Evaluation of retinal nerve fiber layer (RNFL) thickness change (µm), using the average RNFL thickness values measured using Spectral Domain Optical Coherence Tomography (SD-OCT). The change in thickness (µm) will be calculated between the time points described.
Ganglion cell layer thickness change | Baseline, 6 months, 12 months
  Evaluation of ganglion cell layer (GCL+) thickness. This GCL+ thickness is measured using the values for the average ganglion cell layer and inner plexiform layer thickness of the retina (value called "Average GCL + IPL thickness") obtained by Spectral Domain Optical Coherence Tomography (SD-OCT). The change in thickness (µm) will be calculated between the time points described.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Durr, MD, FRCSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Banitt M. Evaluation and management of glaucoma after keratoprosthesis. Curr Opin Ophthalmol. 2011 Mar;22(2):133-6. doi: 10.1097/ICU.0b013e328343723d. PMID 21191292
- [Background] Saheb H, Ahmed II. Micro-invasive glaucoma surgery: current perspectives and future directions. Curr Opin Ophthalmol. 2012 Mar;23(2):96-104. doi: 10.1097/ICU.0b013e32834ff1e7. PMID 22249233
- [Background] Lavia C, Dallorto L, Maule M, Ceccarelli M, Fea AM. Minimally-invasive glaucoma surgeries (MIGS) for open angle glaucoma: A systematic review and meta-analysis. PLoS One. 2017 Aug 29;12(8):e0183142. doi: 10.1371/journal.pone.0183142. eCollection 2017. PMID 28850575
- [Background] Chatzara A, Chronopoulou I, Theodossiadis G, Theodossiadis P, Chatziralli I. XEN Implant for Glaucoma Treatment: A Review of the Literature. Semin Ophthalmol. 2019;34(2):93-97. doi: 10.1080/08820538.2019.1581820. Epub 2019 Feb 21. PMID 30789072
- [Background] Chan HHL, Kong YXG. Glaucoma surgery and induced astigmatism: a systematic review. Eye Vis (Lond). 2017 Nov 17;4:27. doi: 10.1186/s40662-017-0090-x. eCollection 2017. PMID 29177182
- [Background] Pakravan M, Alvani A, Esfandiari H, Ghahari E, Yaseri M. Post-trabeculectomy ocular biometric changes. Clin Exp Optom. 2017 Mar;100(2):128-132. doi: 10.1111/cxo.12477. Epub 2016 Sep 29. PMID 27686794
- [Background] Koivusalo R, Valimaki J. Effect of glaucoma drainage implant surgery on corneal topography: a prospective study. Acta Ophthalmol. 2020 May;98(3):305-309. doi: 10.1111/aos.14247. Epub 2019 Sep 8. PMID 31495070
- [Background] Miraftabi A, Lotfi M, Nilforushan N, Abdolalizadeh P, Jafari S. Ocular biometric changes after Ahmed glaucoma valve implantation. Eur J Ophthalmol. 2021 Jan;31(1):120-124. doi: 10.1177/1120672119889528. Epub 2019 Nov 21. PMID 31752527